CLINICAL TRIAL: NCT07060833
Title: The Use of Bubble Continuous Positive Airway Pressure in Premature Infants: Acoustics as a Metric of Effective Pressure Delivery
Brief Title: Acoustics as a Metric of Airway Pressure in Premature Infants Using Bubble Continuous Positive Airway Pressure
Acronym: Bubble CPAP
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Wissam Shalish, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2025-10708
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Preterm Infant
Keywords: Bubble CPAP; Airflow; Neonatal Intensive Care; Respiratory acoustics; Acoustic monitoring; Airway pressure monitoring; Bubbling sounds
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phase I: 15 preterm infants on Bubble Continuous Positive Airway Pressure (bCPAP): Group 1 will consist of 15 preterm infants on bCPAP in whom the external bubble CPAP sounds and the pressures from the CPAP system itself will be recorded for 3 hours. To do so, we will use a standard microphone placed on the water tank and an external pressure transducer inserted into the expiratory limb of the bubble CPAP circuit.
  Interventions: Device: External pressure transducer; Device: Standard microphone
- Phase II: 15 preterm infants on Bubble Continuous Positive Airway Pressure (bCPAP): Group 2 will consist of 15 preterm infants on bCPAP in whom the external bubble CPAP sounds and the pressures from the CPAP system itself will be recorded. To do so, we will use a standard microphone placed on the water tank and a pressure transducer inserted into the expiratory limb of the bubble CPAP circuit. In addition, the internal bubble CPAP sound and pressure transmitted to the infant's lungs will be measured. For these, a wireless acoustic sensor will be secured on the infant's suprasternal notch to capture transmitted CPAP sounds, and an internal pressure transducer will be inserted from the infant's mouth into the nasopharynx to record the pressure delivered in the airway. Data will be recorded for 3 hours.
  Interventions: Device: External pressure transducer; Device: Standard microphone; Device: Wireless acoustic sensor; Device: Internal pressure transducer

INTERVENTIONS:
Device: External pressure transducer — The delivered CPAP pressure will be measured using an ultra-thin, multi-use catheter pressure transducer inserted into a port in the expiratory limb of the bubble CPAP circuit.
  Other Names: External catheter pressure transducer (Millar Mikro-tip ® SPR-524, 3.5F Single straight, Texas)
Device: Standard microphone — The bubble sound of the water tank will be collected with a standard condenser microphone directly affixed to the pole holding the water tank, with a secure clip.
  Other Names: Lavalier condenser microphone, Tosuny
Device: Wireless acoustic sensor — The wireless acoustic sensor contains a dual microphone capable of capturing target sounds as well as ambient noise. The frequencies associated with ambient noise will be subtracted to maximize the signal-to-noise ratio of the bubble sound waveform. The wireless sensor will be placed on the suprasternal notch of the infant for monitoring the bubble sounds transmitted to the lungs and secured using a silicone-based tape approved for use in neonates. Data will be transmitted in real-time to a research-dedicated tablet using the Bluetooth Communication Controller and stored for future analysis.
  Groups: Phase II: 15 preterm infants on Bubble Continuous Positive Airway Pressure (bCPAP)
Device: Internal pressure transducer — The transmitted CPAP pressure will be measured using an ultra-thin, single-use catheter pressure transducer inserted through the mouth to the level of the infant's nasopharynx. The data will be acquired with a sampling rate of 10kHz and stored for later analysis.
  Groups: Phase II: 15 preterm infants on Bubble Continuous Positive Airway Pressure (bCPAP)

SUMMARY:
This is an observational, proof-of-concept, feasibility study where 30 preterm infants on bubble CPAP with gestational age < 32+0 weeks will be recruited from the neonatal intensive care unit (NICU) at the Montreal Children's Hospital.

The study's main goals are:

1. To determine the relationship between ambient bubbling sounds and delivered pressures in preterm infants on bCPAP.
2. To determine the relationship between transmitted bubbling sounds and airway pressures transmitted to the lungs of preterm infants on bCPAP.
3. To develop models to predict delivered and transmitted bCPAP pressures from the acoustic properties of bubbling sounds.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) is an essential, non-invasive therapy for treating various respiratory conditions in the Neonatal Intensive Care Units (NICU). CPAP is an effective treatment for respiratory distress syndrome, apneas, or after extubation, exerting its physiological benefits by maintaining upper airway patency and functional residual capacity. Bubble CPAP (bCPAP) is the most widely used CPAP due to its low cost and ease of use. It consists of an inspiratory tube carrying heated and humidified air, a nasal interface, and an expiratory tube immersed in a water chamber. The generation of bubbles in the water chamber by exhaled gas creates low amplitude and high-frequency pressure oscillations that are transmitted back to the chest. Successful CPAP requires constant transmission of the pressure via an unobstructed circuit. However, this is difficult to achieve in practice due to inadequate interface, leaks from an open mouth, and obstructed airway. As a result, bCPAP requires frequent manual checks by nurses and respiratory therapists to ensure that the circuit is secure and unobstructed.

As a proposed solution, bCPAP sounds heard in the patient room or upon auscultation are routinely used to assess the effectiveness of CPAP therapy. This sound can be heard both from the water tank creating the vibrations and during auscultation with a stethoscope, as the sound vibration is transmitted to the neonatal lungs. In the current era of digital technology, acoustic sounds can be converted to electronic signals for further processing and analysis.

We hypothesize that continuous recording and analysis of bCPAP sounds could be used as a proxy for real-time objective monitoring of the pressure transmitted to infants' lungs.

ELIGIBILITY:
Inclusion Criteria:

* Infants on bCPAP with gestational age < 32+0 weeks
* Postmenstrual age between 28+0 and 36+6 weeks at the time of the study
* Postnatal age greater than 168 hours (7 days) at the time of the study
* On the bubble CPAP device with binasal prongs at the time of the study
* Receiving bubble CPAP levels of 5 to 7 cm H2O with gas flows between 6L/min and 10L/min at the time of the study

Exclusion Criteria:

* Infants with known major congenital anomalies
* Infants with known congenital heart disorders
* Infants with known neuromuscular disease
* Infants receiving ventilator-derived CPAP at the time of the study
* Infants receiving CPAP via a nasal mask interface at the time of the study
* Infants receiving inotropes, narcotics or sedative agents at the time of the study
* Infants deemed clinically unstable for the study by the attending neonatologist

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to the neonatal intensive care unit at the Montreal Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pressure | 3 hours
  The mean pressure and the standard deviation of the pressure will be computed for each segment.
External bubble CPAP sounds | 3 hours
  Two metrics will be computed:
  1. The root mean square (RMS)
  2. The power contained between a pre-determined range within each segment; We will determine the range that contains 80% of the signal power, in order to minimize other noises from bubble CPAP signal.
Internal bubble CPAP sounds | 3 hours
  1. We will apply biomedical signal processing methods to separate the bubbling sounds from breathing sounds. Then, RMS and power will be computed.
  2. We will use the Pearson correlation coefficient to compute the relationship between bubbling sound and pressure metrics. We will evaluate the linear regression models to identify the combination of sound metrics and covariates with the highest predictive accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Shalish, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No